CLINICAL TRIAL: NCT05145751
Title: SARS CoV-2 Infection and Simple Inflammatory Biomarkers.
Brief Title: SARS CoV-2 Infection and Inflammatory Biomarkers
Status: Completed | Type: Observational
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Elena Arnaoutoglou, Professor of Anesthesiology, University of Thessaly
Other Study IDs: 46937
Record Dates: First submitted 2021-12-02; First posted 2021-12-06 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: COVID-19; Inflammation
Keywords: COVID-19; Biomarkers; Inflammation
MeSH Terms: conditions — COVID-19; Inflammation | interventions — Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 infection: Consecutive patients with polymerase chain reaction (PCR) confirmed SARS CoV-2 infection
  Interventions: Other: Simple inflammatory biomarkers measurement

INTERVENTIONS:
Other: Simple inflammatory biomarkers measurement — In patients with polymerase chain reaction (PCR) confirmed SARS CoV-2 infection the values of simple inflammatory biomarkers such NLR will be measured
  Other Names: Consecutive patients with polymerase chain reaction (PCR) confirmed SARS CoV-2 infection

SUMMARY:
Early research suggests that inflammation plays a key role in the development of SARS CoV-2 infection. The immune response to respiratory infection is characterized by an influx of neutrophils to the lungs. This study ought to investigate the association of simple biomarkers such as NLR and PLR with the clinical outcome in SARS CoV-2 infection patients.

DETAILED DESCRIPTION:
Early research suggests that inflammation plays a key role in the development of SARS CoV-2 infection. The immune response to respiratory infection is characterized by an influx of neutrophils to the lungs. Moreover, previous studies have demonstrated that a sustained release of anti-inflammatory cytokines may lead to high levels of circulating neutrophils and lymphocytes' apoptosis with subsequent lymphopenia and immune response imbalance. Therefore, circulating biomarkers that represent inflammation and immune status could serve as potential predictors for the prognosis of SARS CoV-2 patients. The neutrophil to lymphocyte ratio (NLR) and platelet to lymphocyte ratio (PLR) are cheap and simply calculated biomarkers which have been identified as markers of systemic inflammation, severity of the disease and prognosis in several patient populations.

This study ought to investigate the association of simple biomarkers such as NLR and PLR with the clinical outcome in SARS CoV-2 infection patients.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with polymerase chain reaction (PCR) confirmed SARS CoV-2 infection

Exclusion Criteria:

* Patients aged<18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with SARS CoV-2 infection who were treated by the Department of Respiratory Medicine in the UHL will be done. The subjects will be followed from admission to the hospital and up until discharge, transfer to the ICU or death
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Outcome | 1 year
  Outcome after COVID-19 infection

CONTACTS AND LOCATIONS:
Overall Officials: Eleni Arnaoutoglou, M.D., Ph.D., Study Chair — Study Chair
Locations (1):
- Univeristy of Thessaly, Larissa, Thessaly, Greece